CLINICAL TRIAL: NCT05198141
Title: Evaluation of Different Doses of Aromatase Inhibitor Letrozole for the Treatment of Ectopic Pregnancy
Brief Title: Evaluation of Different Doses of Letrozole in Ectopic Pregnancy
Acronym: letrezole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed Ali Alabiad, MD, Principal Investigator, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LETROZOLE ON ECTOPIC PREGNANCY
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Ectopic Pregnancy
Keywords: LETREZOLE; Ectopic pregnancy; Induced abortion
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group I (GI) (Active Comparator): Patients who were undergoing surgical treatment
  Interventions: Procedure: laparoscopic salpingectomy
- low dose letrozole group II (GII) (Experimental): patients who were medically treated with 5 mg of letrozole
  Interventions: Drug: Letrozole tablets
- High dose letrozole group (GIII) (Experimental): patients who were medically treated with 10 mg of letrozole using
  Interventions: Drug: Letrozole tablets

INTERVENTIONS:
Drug: Letrozole tablets — GI: Patients who were undergoing laparoscopic salpingectomy GII: patients who medically treated with 5 mg d-1 of letrozole using two tablets (2.5 mg of Femara) every day for 10 d GIII patients who medically treated with 10 mg d-1 of letrozole using four tablets (2.5 mg of Femara) every day for 10 d (group III)
  Other Names: Femara
  Arms: High dose letrozole group (GIII); low dose letrozole group II (GII)
Procedure: laparoscopic salpingectomy — laparoscopic salpingectomy
  Arms: Control group I (GI)

SUMMARY:
The utilization of letrozole at a daily dose of 10 mg for medical treatment of ectopic pregnancy considerably has a high success rate without imposing any serious side effects compared to daily 5mg letrozole.

DETAILED DESCRIPTION:
Letrozole, an aromatase inhibitor, has recently been introduced as favorable medical treatment for ectopic pregnancy. We aimed at evaluating the effects of different doses of letrozole for induction of abortion Sixty patients with undisturbed ectopic pregnancy were classified into three equal groups. Group I: The control group that contained women who were undergoing laparoscopic salpingectomy, Group II: Patients who received letrozole (5 mg d-1) for 10 d, and Group III: Patients who received letrozole (10 mg d-1) for 10 d. After that, the human chorionic gonadotropin (β-hCG) levels were determined for the first day and after 11 d of treating. letrozole (10 mg d-1) markedly reduced the receptors of estrogen and progesterone, and subsequent vascular endothelial growth factor signals, resulting in marked apoptosis in the placenta tissue. The utilization of letrozole at a dose of 10 mg d-1 for inducement of abortion typically results in a substantial high-successful rate without any severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ectopic pregnancy was by
* Absence of an intrauterine gestational sac on vaginal ultrasound Coupled with
* β-hCG titers beyond the discrimination zone of at least 2,000 milli-International units (mIU/m).

Exclusion Criteria:

* Patients had contraindications for letrozole
* Patients with any systemic disease ( diabetes, hypertension, ....)
* Patients with b-hCG levels >3,000 mIU/mL
* Patients with hemoglobin level <10 g/dL,
* Patients with platelets count <150,000/mL,
* Patients with elevated liver enzymes,
* Patients with elevated blood urea, or serum creatinine
* The presence of a fetal heartbeat in a gestational sac detected outside the uterine cavity

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
β-hCG level | The β-hCG levels were assessed on the 1st of treatment
  A quantitative human chorionic gonadotropin
β-hCG level | The β-hCG levels were assessed on the 11th day of treatment
  A quantitative human chorionic gonadotropin

SECONDARY OUTCOMES:
Complete blood count (CBC) | Assessed on the 1st day of treatment
  Complete blood count
Alanine Amino Transferase (ALT) | Assessed on the 1st and 11th day of treatment
  Liver enzyme
Aspartate aminotransferase (AST) | Assessed on the 1st and 11th day of treatment
  Liver enzyme
Serum creatinine | Assessed on the 1st and 11th day of treatment
  Renal function test
Blood urea | Assessed on the 1st and 11th day of treatment
  Renal function test
Complete blood count (CBC) | Assessed on the 11th day of treatment
  Complete blood count
Alanine Amino Transferase (ALT) | Assessed on the 11th day of treatment
  Liver enzyme
Aspartate aminotransferase (AST) | Assessed on the 11th day of treatment
  Liver enzyme
Serum creatinine | Assessed on the 11th day of treatment
  Renal function test
Blood urea | Assessed on the 11th day of treatment
  Renal function test

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Heraiz, MD, Principal Investigator — Zagazig University
Locations (1):
- Mohamed ALI Alabiad, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Table Statistical analysis Master sheet raw data (excel sheet)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: the data will become available after one month from the approval and will be available for three months
Access Criteria: you can send a Data request email to Dr: Mohamed at drno99@yahoo.com

REFERENCES:
- Available data/document: Study Protocol — http://www.staffdata.zu.edu.eg/ar/ShowData/23528 — you can send a Data request e-mail to Dr Mohamed at drno99@yahoo.com
- Available data/document: Statistical Analysis Plan: drno99@yahoo.com — http://www.staffdata.zu.edu.eg/ar/ShowData/23528 — you can send a Data request e-mail to Dr Mohamed at drno99@yahoo.com
- Available data/document: Informed Consent Form — http://www.staffdata.zu.edu.eg/ar/ShowData/23528 — you can send a Data request e-mail to Dr Mohamed at drno99@yahoo.com
- Available data/document: Individual Participant Data Set — http://www.staffdata.zu.edu.eg/ar/ShowData/23528 — you can send a Data request e-mail to Dr Mohamed at drno99@yahoo.com